CLINICAL TRIAL: NCT05195008
Title: A Phase 1 Randomized, Blinded, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics, With an Open-Label Target Occupancy Study of BIIB113 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics, With Target Occupancy Study of BIIB113 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 276HV101; 2021-002903-36 (EudraCT Number)
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part A [Single Ascending Dose (SAD)]: BIIB113 Cohort 1 (Experimental): Participants aged 18 to 64 years will receive Dose 1 of BIIB113, orally, once daily (QD), on Day 1 of Part A of the study.
  Interventions: Drug: BIIB113
- Part A (SAD): BIIB113 Cohort 2 (Experimental): Participants aged 18 to 64 years will receive Dose 2 of BIIB113, orally, QD, on Day 1 of Part A of the study
  Interventions: Drug: BIIB113
- Part A (SAD): BIIB113 Cohort 3 (Experimental): Participants aged 18 to 64 years will receive Dose 3 of BIIB113, orally, QD, on Day 1 of Part A of the study.
  Interventions: Drug: BIIB113
- Part A (SAD): BIIB113 Cohort 4 (Experimental): Participants aged 18 to 64 years will receive Dose 4 of BIIB113, orally, QD, on Day 1 of Part A of the study.
  Interventions: Drug: BIIB113
- Part A (SAD): BIIB113 Cohort 5 (Experimental): Participants aged 18 to 64 years will receive Dose 5 of BIIB113, orally, QD, on Day 1 of Part A of the study
  Interventions: Drug: BIIB113
- Part A (SAD): BIIB113-Matching Placebo (Cohorts 1-5) (Placebo Comparator): Participants aged 18 to 64 years will receive BIIB113-matching placebo, orally, QD, on Day 1 of Part A of the study.
  Interventions: Drug: BIIB113-Matching Placebo
- Part B [Multiple Ascending Dose (MAD)]: BIIB113 Cohort 6 (Experimental): Participants aged 18 to 64 years will receive Dose 3 of BIIB113, orally, QD, up to Day 14 of Part B of the study.
  Interventions: Drug: BIIB113
- Part B (MAD): BIIB113 Cohort 7 (Experimental): Participants aged 18 to 64 years will receive Dose 4 of BIIB113, orally, QD, on Days 1 to 14 of Part B of the study.
  Interventions: Drug: BIIB113
- Part B (MAD): BIIB113 Cohort 8 (Experimental): Participants aged 18 to 64 years will receive Dose 6 of BIIB113, orally, QD, on Days 1 to 14 of Part B of the study.
  Interventions: Drug: BIIB113
- Part B (MAD): BIIB113 Cohort 9 (Placebo Comparator): Participants aged 65 to 75 years will receive BIIB113, orally, QD, on Days 1 to 14 of Part B of the study. The calculated dose level will be adaptive by design based on review of the safety, tolerability, and PK data from Cohorts 1 to 7.
  Interventions: Drug: BIIB113
- Part B (MAD): BIIB113-Matching Placebo (Cohorts 6 to 9) (Placebo Comparator): Participants aged 18 to 75 will receive BIIB113-matching placebo, orally, QD, on Days 1 to 14 of Part B of the study.
  Interventions: Drug: BIIB113-Matching Placebo
- Part C (OGA-PET SAD): BIIB113 (Experimental): Participants aged 20 to 64 will receive single dose of BIIB113, orally, QD, on Day 1 of Part C of the study, followed by a radiotracer specific to OGA ([11^C]BIO-1819578), on Days 1 to 4 of Part C of the study.
  Interventions: Drug: BIIB113; Drug: 11^C]BIO-1819578
- Part C (OGA-PET MAD): BIIB113 (Experimental): Participants aged 20 to 64 years will receive multiple doses of BIIB113, orally, QD, on Days 1 to 14 of Part C of the study, followed by a radiotracer specific to OGA ([11^C]BIO-1819578) on Day 1 and either of Day 15, Day 16 or Day 17 of Part C of the study.
  Interventions: Drug: BIIB113; Drug: 11^C]BIO-1819578

INTERVENTIONS:
Drug: BIIB113 — Administered as specified in the treatment arm.
  Arms: Part A (SAD): BIIB113 Cohort 2; Part A (SAD): BIIB113 Cohort 3; Part A (SAD): BIIB113 Cohort 4; Part A (SAD): BIIB113 Cohort 5; Part A [Single Ascending Dose (SAD)]: BIIB113 Cohort 1; Part B (MAD): BIIB113 Cohort 7; Part B (MAD): BIIB113 Cohort 8; Part B (MAD): BIIB113 Cohort 9; Part B [Multiple Ascending Dose (MAD)]: BIIB113 Cohort 6; Part C (OGA-PET MAD): BIIB113; Part C (OGA-PET SAD): BIIB113
Drug: BIIB113-Matching Placebo — Administered as specified in the treatment arm.
  Arms: Part A (SAD): BIIB113-Matching Placebo (Cohorts 1-5); Part B (MAD): BIIB113-Matching Placebo (Cohorts 6 to 9)
Drug: 11^C]BIO-1819578 — Administered as specified in the treatment arm.
  Arms: Part C (OGA-PET MAD): BIIB113; Part C (OGA-PET SAD): BIIB113

SUMMARY:
Parts A and B: The primary objective of this study is to evaluate the safety and tolerability of single and multiple ascending oral doses of BIIB113 in healthy participants. The secondary objectives of this study are to evaluate the single and multiple oral dose pharmacokinetic (PK) profile of BIIB113 in healthy participants and to evaluate the effect of food on the single oral dose of BIIB113 in healthy participants of Part A cohort 3.

Part C: The primary objectives of this study are to evaluate the safety and tolerability of single and multiple ascending oral doses of BIIB113 in healthy participants and to determine target occupancy (TO) as measured by O-GlcNAcase-Positron Emission Tomography (OGA-PET) of single and multiple oral doses of BIIB113 in healthy participants.

DETAILED DESCRIPTION:
BIIB113 is a small molecule inhibitor of OGA being evaluated in Alzheimer's disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Female or infertile/vasectomized males aged 18 to 64 years (Parts A and B), 20 to 64 years (Part C), or 65 to 75 years (Part B Dose 7Cohort 9 only), inclusive, at the time of informed consent
* Have a body mass index between 18 and 32 kilograms per square meter (kg/m^2), inclusive, at screening
* Weight ≥50 kilograms (kg) at screening
* Negative Polymerase Chain Reaction (PCR) test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) within 5 days of Day -1 prior to randomization

Key Exclusion Criteria:

* History or positive test result at Screening for Human Immunodeficiency Virus (HIV)
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia), as determined by the investigator, within 90 days prior to screening or between screening and Day -1
* History of severe allergic or anaphylactic reactions, or of any allergic reactions that in the opinion of the investigator are likely to be exacerbated by any component of the study treatment
* History of systemic hypersensitivity reaction to BIIB113 or the excipients contained in the formulation, and if appropriate, any diagnostic agents to be administered during the study
* Has suicidal ideation with some intent to act within 6 months prior to the start of screening, per the investigator's clinical judgment or based on the C-SSRS, corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) for suicidal ideation on the C-SSRS, or a history of suicidal behaviour within one year prior to the start of screening.
* Any condition affecting study treatment absorption (e.g., gastrectomy)
* Previous exposure to an OGA inhibitor
* Current enrolment in any other drug, biologic, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 90 days (6 months for biologics) prior to Day -1, or 5 half-lives of the agent, whichever is longer
* For Part C only: Previously undergone PET scans for research purposes

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Parts A, B and C: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Part A: Up to 54 days; Part B: Up to 53 days; Part C: Up to 71 days (SAD); Up to 85 days (MAD)
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death; in the view of the investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or is a medically important event.
Parts A, B and C: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Parameters, Vital Signs, and 12-Lead Electrocardiogram (ECG) | Part A: Baseline up to 54 days; Part B: Baseline up to 53 days; Part C: Baseline up to 71 days (SAD), Baseline up to 85 days (MAD)
Parts A, B and C: Number of Participants With Change in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Part A: Up to 54 days; Part B: Up to 53 days; Part C: Up to 71 days (SAD); Up to 85 days (MAD)
  C-SSRS is used to assess the suicidality of participants during the study. The assessment includes "yes" or "no" responses for 5 questions each, related to suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Numeric ratings are provided for severity of ideation, from 1 to 5, with 5 being the most severe.
Part C: Percent O-GlcNAcase-Positron Emission Tomography (OGA PET) Target Engagement/Occupancy (TO) as a Function of Dose and Time | Up to Day 4 (SAD); Up to Day 17 (MAD)

SECONDARY OUTCOMES:
Parts A and B: Area Under the Concentration-Time Curve From Time Zero to Time of the Last Measurable Concentration (AUClast) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC∞) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Area Under the Plasma Concentration-Time Curve Within a Dosing Interval (AUCtau) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Maximum Observed Concentration (Cmax) for BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Trough Concentration (Ctrough) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Time to Maximum Observed Concentration (Tmax) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Terminal Elimination Half-Life (t½) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  t1/2 is the time measured for the plasma concentration to decrease by one half. The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Apparent Total Body Clearance (CL/F) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. If the bioavailability (F) of a dose is assumed to be 100% or equivalently, that clearance is the apparent clearance (CL/F) when the ratio of clearance to bioavailability is assumed to be constant.
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  Volume of distribution is defined as the apparent volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Accumulation Ratio (AR) of BIIB113 | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Amount of BIIB113 Excreted in Urine (Aeu) | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.
Parts A and B: Percentage of BIIB113 Excreted in Urine (%fe) | Part A: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part B: Pre-dose and at multiple timepoints post-dose on Days 1 to 15
  The parameter will be assessed under fed conditions for Part A Cohort 3.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- Karolinska Comprehensive Cancer Center - Studieenheten, Flemingsberg, Stockholm County, Sweden
- United Kingdom (2):
  - Hammersmith Medicine Research, London, Brent
  - Medicines Evaluation Unit, Wythenshawe, Manchester

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/